CLINICAL TRIAL: NCT01012622
Title: An Open-label Prospective Trial to Evaluate Functional Outcomes of OROS Methylphenidate in Children With ADHD (FOSCO)
Brief Title: An Efficacy and Safety Study of Osmotic Release Oral System (OROS) Methylphenidate in Participants With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015481; CON-KOR-4020
Record Dates: First submitted 2009-11-05; First posted 2009-11-13 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate Hydrochloride
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OROS Methylphenidate Hydrochloride (Experimental)
  Interventions: Drug: Osmotic Release Oral System (OROS) Methylphenidate Hydrochloride

INTERVENTIONS:
Drug: Osmotic Release Oral System (OROS) Methylphenidate Hydrochloride — OROS methylphenidate hydrochloride (HCL) will be given orally once daily at an initial dose of 18 milligram (mg) for participants below 30 Kilogram (kg) and 27 mg for those over 30 kg of body weight. The dose will be increased by 9 mg or 18 mg every week for up to Week 8, followed by a maximum maintenance dose of 54 mg orally once daily up to Week 12 during which the dose can be decreased by 9 mg depending on tolerability.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Osmotic Release Oral System (OROS) methylphenidate in participants with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This is an open-label (all people involved know the identity of the intervention), single arm, multicenter (when more than one hospital or medical school team work on a medical research study), prospective study (study following participants forward in time) to evaluate the efficacy and safety of OROS methylphenidate in participants with ADHD (behavior disorder originating in childhood in which the essential features are signs of developmentally inappropriate inattention, impulsivity, and hyperactivity). The study duration will be of 12 weeks per participant, which is divided into 2 parts Screening (within 14 days before study commences on Day -1) and treatment (8 weeks and will include titration period [from the initiation of the study treatment to determination of the individual's maintenance dose] and maintenance period [at least 4 weeks after determination of maintenance dose]). Participants will receive initial dose depending on their body weight. OROS methylphenidate hydrochloride (HCL) will be given orally once daily at an initial dose of 18 milligram (mg) for participants below 30 kilogram (kg) and 27 mg for those over 30 kg of body weight. The dose will be increased by 9 mg or 18 mg every week for up to Week 8, followed by a maximum maintenance dose of 54 mg orally once daily up to Week 12 during which the dose can be decreased by 9 mg depending on tolerability. Efficacy will be evaluated by Korean Version, ADHD Rating Scale (K-ARS) total score and Clinical Global Impression)-Severity / Impression rating scale CGI-S/I. Participants safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily provided informed consent to participate in the study
* Participants with written informed consent to participate in the study voluntarily by caregivers/legal representatives
* Participants who were capable to follow the study visit schedule well and their parents/caregivers who were willing to complete the assessments specified in the protocol and were capable to complete them
* Participant and his/her parent/guardian able to understand the study participation and to request withdrawal from the study voluntarily at any time
* Participants who were satisfied in diagnosis of Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) Attention Deficit Hyperactivity Disorder (ADHD) and determined to require drug therapy

Exclusion Criteria:

* Participants who have known hypersensitivity (altered reactivity to an antigen, which can result in pathologic reactions upon subsequent exposure to that particular antigen) to methylphenidate HCL
* Participants who have significant suicidal ideation
* Participants with mental retardation
* Participants who meet DSM-IV diagnostic criteria for current major depressive disorder or anxiety disorder requiring drug therapy
* Participants who have abnormalities in the Electrocardiography (ECG) or show clinically significant abnormalities of laboratory results, including serum chemistries and hematology

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- [Derived] Kim BN, Cummins TD, Kim JW, Bellgrove MA, Hong SB, Song SH, Shin MS, Cho SC, Kim JH, Son JW, Shin YM, Chung US, Han DH. Val/Val genotype of brain-derived neurotrophic factor (BDNF) Val(6)(6)Met polymorphism is associated with a better response to OROS-MPH in Korean ADHD children. Int J Neuropsychopharmacol. 2011 Nov;14(10):1399-410. doi: 10.1017/S146114571100099X. Epub 2011 Jun 28. PMID 21733227

RESULTS

PARTICIPANT FLOW:
Groups:
- Osmotic Release Oral System (OROS) Methylphenidate HCL: OROS methylphenidate hydrochloride (HCL) was given orally once daily at an initial dose of 18 milligram (mg) for participants below 30 Kilogram (kg) and 27 mg for those over 30 kg of body weight. The dose was increased by 9 mg or 18 mg every week for up to Week 8, followed by a maximum maintenance dose of 54 mg orally once daily up to Week 12 during which the dose can be decreased by 9 mg depending on tolerability.
Period: Overall Study
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Started | 142
Completed | 111
Not Completed | 31
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 7
Not completed — non-compliance with the drug | 9
Not completed — Other | 1
Not completed — screening failure | 1
Not completed — withdrawal of consent by a parent | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who took at least one dose of study drug.
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 112

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Korean Version of the Attention-Deficit Hyperactivity Disorder (K-ADHD) Rating Scale (K-ARS) Total Score at Week 12
Description: K-ARS measures the 18 symptoms based on Diagnostic and Statistical Manual of Mental Disorders-forth edition (DSM-IV 1994). Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often), whereas the rating of 2 points or more was regarded as abnormal. Total scores range from 0 (no symptoms) to 54 (highly symptomatic), higher score indicates worsening of condition.
Time Frame: Baseline and Week 12
Population: Intention-to-treat (ITT) population included participants who received the study drug at least once and had the primary efficacy endpoint data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 134
units on a scale
  Baseline | 33.37 (8.67)
  Change at Week 12 | -20.43 (10.42)

2. Primary Outcome: Number of Participants With Response Based on K-ARS Total Score at Week 12
Description: Response is defined as at least 25 percent (%) decrease in total score of K-ARS compared to baseline. K-ARS measures the 18 symptoms based on DSM-IV (1994). Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often), whereas the rating of 2 points or more was regarded as abnormal. Total scores range from 0 (no symptoms) to 54 (highly symptomatic), higher score indicates worsening of condition.
Time Frame: Week 12
Population: ITT population included participants who received the study drug at least once and had the primary efficacy endpoint data available. "N" (Number of Participants Analyzed) represents number of participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 127
participants | 118

3. Primary Outcome: Number of Participants With Remission Based on K-ARS Total Score and Clinical Global Impression - Improvement (CGI-I) Scale Score at Week 12
Description: Remission is defined by all of the following criteria; 1) K-ARS Total score of 18 or less. 2) "Very much improved" or "Much improved" in CGI-I. K-ARS total score ranges from 0 (no symptoms) to 54 (highly symptomatic), higher score indicates worsening of condition. CGI-I is a 7-point scale ranging from 1 to 7, where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse, higher score indicates worsening of condition.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 127
participants | 99

4. Secondary Outcome: Change From Baseline in Child Health and Illness Profile-Child Edition (CHIP) Total Score and 5 Sub-domains Score at Week 12
Description: CHIP was designed to assess the physical, psychological health conditions and functional well-being of children. The instrument has sub-domains such satisfaction (11 items) ranges from 0 to 44, stability (22 items) ranges from 0 to 88, elasticity (19 items) ranges from 0 to 76, risk aversion (14 items) ranges from 0 to 56, achievement (10 items) ranges from 0 to 40. Good health is in the range from 44 to 56 points for all sub-domains. A score of 43 or below indicates poor health in that domain. A score of 57 or higher indicates excellent health. The total score is an average of the scores for the 5 domains and ranges from 0 to 304. Higher total score indicates better health.
Time Frame: Baseline and Week 12
Population: ITT population included participants who took study drug at least once and had primary efficacy endpoint data available. Last Observation Carried Forward (LOCF) method was used. "n" signifies participants who were evaluated for each specified category for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 134
units on a scale
  Total Score:Baseline (n=126) | 207.85 (26.62)
  Total Score:Change at Week 12 (n=126) | 18.08 (22.54)
  Satisfaction:Baseline (n=132) | 26.17 (7.20)
  Satisfaction:Change at Week 12 (n=132) | 2.27 (5.89)
  Stability:Baseline (n=129) | 82.13 (11.18)
  Stability:Change at Week 12 (n=129) | 4.47 (10.87)
  Elasticity:Baseline (n=132) | 38.30 (8.22)
  Elasticity:Change at Week 12 (n=132) | 2.53 (7.10)
  Risk aversion:Baseline (n=132) | 40.67 (7.91)
  Risk aversion:Change at Week 12 (n=132) | 5.73 (7.27)
  Achievement:Baseline (n=133) | 21.00 (6.16)
  Achievement:Change at Week 12 (n=133) | 2.45 (5.07)

5. Secondary Outcome: Change From Baseline in Visual Selective Attention Subtest of Comprehensive Attention Test (CAT) Total Score at Week 12
Description: CAT was developed to properly reflect brain function in childhood. It provided measurement of simple visual selective attention in terms of omission (number of missing response to target stimulus [0-150], higher score indicate greater omission), false alarm (number of response to non-target stimulus [0-150], higher score indicate greater false alarm), response mean (average time spent to response to target stimulus [200-1100, low score means faster response to target stimulus]), Response (consistency of response time to target stimulus [30-650, Low score means good consistency of response]).
Time Frame: Baseline and Week 12
Population: ITT population included participants who received the study drug at least once and had the primary efficacy endpoint data available. LOCF method was used. "N" (Number of Participants Analyzed) represents number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 118
units on a scale
  Omission:Baseline | 8.79 (15.77)
  Omission:Change at Week 12 | -4.53 (17.94)
  False alarm:Baseline | 17.42 (18.48)
  False alarm:Change at Week 12 | -5.03 (13.43)
  Response mean:Baseline | 501.32 (130.80)
  Response mean:Change at Week 12 | -37.41 (110.34)
  Response:Baseline | 201.05 (105.78)
  Response:Change at Week 12 | -48.36 (111.02)

6. Secondary Outcome: Change From Baseline in Auditory Selective Attention Subtest of Comprehensive Attention Test (CAT) Total Score at Week 12
Description: CAT was developed to properly reflect brain function in childhood. It provided measurement of simple auditory selective attention in terms of omission (number of missing response to target stimulus [0-150], higher score indicate greater omission), false alarm (number of response to non-target stimulus [0-150], higher score indicate greater false alarm), response mean (average time spent to response to target stimulus [200-1100, low score means faster response to target stimulus]), Response (consistency of response time to target stimulus [30-650, Low score means good consistency of response]).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 118
units on a scale
  Omission:Baseline | 10.31 (16.52)
  Omission:Change at Week 12 | -6.27 (15.88)
  False alarm:Baseline | 12.07 (14.41)
  False alarm:Change at Week 12 | -3.61 (11.86)
  Response mean:Baseline | 623.95 (188.38)
  Response mean:Change at Week 12 | -55.34 (155.36)
  Response:Baseline | 265.69 (108.76)
  Response:Change at Week 12 | -63.76 (114.15)

7. Secondary Outcome: Change From Baseline in Inhibition-Sustained Attention Subtest of Comprehensive Attention Test (CAT) Total Score at Week 12
Description: CAT was developed to properly reflect brain function in childhood. It provided measurement of simple inhibition-sustained attention in terms of omission(number of missing response to target stimulus [0-150], higher score indicate greater omission), false alarm(number of response to non-target stimulus [0-150], higher score indicate greater false alarm), response mean (average time spent to response to target stimulus [200-1100, low score means faster response to target stimulus]), Response (consistency of response time to target stimulus [30-650, Low score means good consistency of response]).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 119
units on a scale
  Omission:Baseline | 35.78 (46.91)
  Omission:Change at Week 12 | -20.39 (45.40)
  False alarm:Baseline | 27.73 (15.58)
  False alarm:Change at Week 12 | -7.54 (14.19)
  Response mean:Baseline | 576.55 (147.13)
  Response mean:Change at Week 12 | -34.44 (140.43)
  Response:Baseline | 273.78 (121.94)
  Response:Change at Week 12 | -66.85 (127.13)

8. Secondary Outcome: Change From Baseline in Interference-Selective Attention Subtest of Comprehensive Attention Test (CAT) Total Score at Week 12
Description: CAT was developed to properly reflect brain function in childhood. It provided measurement of simple interference-selective attention in terms of omission(number of missing response to target stimulus[0-150], higher score indicate greater omission), false alarm(number of response to non-target stimulus[0-150], higher score indicate greater false alarm), response mean (average time spent to response to target stimulus [200-1100, low score means faster response to target stimulus]), Response (consistency of response time to target stimulus [30-650, Low score means good consistency of response]).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 119
units on a scale
  Omission:Baseline | 20.39 (24.44)
  Omission:Change at Week 12 | -10.83 (20.10)
  False alarm:Baseline | 26.03 (18.30)
  False alarm:Change at Week 12 | -6.14 (16.75)
  Response mean:Baseline | 648.48 (171.84)
  Response mean:Change at Week 12 | -54.35 (134.26)
  Response:Baseline | 276.74 (156.70)
  Response:Change at Week 12 | -72.18 (148.01)

9. Secondary Outcome: Change From Baseline in Divided Attention Subtest of Comprehensive Attention Test (CAT) at Week 12
Description: CAT was developed to properly reflect brain function in childhood. It provided measurement of simple divided attention in terms of omission(number of missing response to target stimulus[0-150], higher score indicate greater omission), false alarm(number of response to non-target stimulus[0-150], higher score indicate greater false alarm), response mean (average time spent to response to target stimulus [200-1100, low score means faster response to target stimulus]), Response (consistency of response time to target stimulus [30-650, Low score means good consistency of response]).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 59
units on a scale
  Omission:Baseline | 16.05 (9.69)
  Omission:Change at Week 12 | -4.07 (10.18)
  False alarm:Baseline | 16.03 (12.36)
  False alarm:Change at Week 12 | -4.73 (9.44)
  Response mean:Baseline | 749.01 (196.66)
  Response mean:Change at Week 12 | -27.14 (186.70)
  Response:Baseline | 349.60 (130.41)
  Response:Change at Week 12 | -43.90 (118.84)

10. Secondary Outcome: Change From Baseline in Working Memory Forward Subtest of Comprehensive Attention Test (CAT) at Week 12
Description: CAT was developed to properly reflect brain function in childhood. The test battery provided a comprehensive measurement of simple visual auditory attention, interventional visual-auditory selective attention, divided attention, continuous attention, and operational memory. Working memory forward was measured in terms of width of space and number of correct responses ranging from 0 to 10. For width of space boxes were presented on the screen and participants remembered the order of presented box. Participants pressed the box using mouse in the forward order. Maximum number that participants correctly memorized box in the screen in the respective order was reported and overall number of times a participant responded correctly was also reported.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 59
correct responses
  Baseline:Number of correct responses | 5.76 (2.34)
  Change at Week 12:Number of correct responses | 0.63 (2.56)
  Baseline:Width of space | 4.46 (1.53)
  Change at Week 12:Width of space | 0.25 (1.78)

11. Secondary Outcome: Change From Baseline in Working Memory Backward Subtest of Comprehensive Attention Test (CAT) at Week 12
Description: CAT was developed to properly reflect brain function in childhood. The test battery provided a comprehensive measurement of simple visual auditory attention, interventional visual-auditory selective attention, divided attention, continuous attention, and operational memory. Working memory forward was measured in terms of width of space and number of correct responses ranging from 0 to 10. For width of space boxes were presented on the screen and participants remembered the order of presented box. Participants pressed the box using mouse in the backward order. Maximum number that participants correctly memorized box in the screen in the respective order was reported and overall number of times a participant responded correctly was also reported.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 59
correct responses
  Baseline:Number of correct responses | 4.22 (2.79)
  Change at Week 12:Number of correct responses | 1.86 (3.02)
  Baseline:Spatial span | 3.63 (2.06)
  Change at Week 12:Spatial span | 1.24 (1.98)

12. Secondary Outcome: Change From Baseline in Academic Performance Rating Scale (APRS) Score at Week 12
Description: APRS scale measures four factors in elementary school children such as learning ability, academic performance, impulse control, and social withdrawal. In particular, it is excellent in assessing drug effect on the academic performance not measured by other scales. Score ranges from 19 to 95, higher score means better academic performance.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 125
units on a scale
  Baseline | 55.46 (12.77)
  Change at Week 12 | 7.40 (9.86)

13. Secondary Outcome: Change From Baseline in Beck Depression Inventory (BDI) Score at Week 12
Description: Beck Depression Inventory (BDI) consisted of 21 items for measuring the subjective severity of depression and emotional, cognitive, motivational, physiological symptoms of depression. Each question has a set of 4 possible answer choices, ranging in intensity, each answer being scored on a scale value of 0 (no symptom) to 3 (the most severe symptom). Accordingly, the total score ranges from 0 (no symptom) to 63 (the most severe symptom) for 21 questions.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 127
units on a scale
  Baseline | 11.69 (7.79)
  Change at Week 12 | -1.89 (6.59)

14. Secondary Outcome: Change From Baseline in Parenting Stress Index (PSI) Total Score at Week 12
Description: Parenting Stress Index (PSI) was designed to assess parent or guardian child-rearing stress index on a 5-rating scale from "never" to "very truly". Out of 30 items, 20 items are scored, being consisted of 8 child characteristics-related stress items; 9 parent-child interaction-related stress items; and 3 achievement expectation-related stress items. A possible total score ranges from 20 to 100; Increase in score indicates higher stress perceived by the parent.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 123
units on a scale
  Baseline | 58.20 (9.33)
  Change at Week 12 | -5.25 (9.01)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression-severity (CGI-S) Score at Week 12
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher change scores indicate worsening.
Time Frame: Baseline and Week 12
Population: ITT population included participants who received the study drug at least once and had the primary efficacy endpoint data available. LOCF method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 134
units on a scale
  Baseline | 5.14 (0.90)
  Change at Week 12 | -2.51 (1.36)

16. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Scale Score at Week 12
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Improved very much, Improved much and Improved a little are defined as improvement and No change, Aggravated a little, Aggravated much and Aggravated very much were defined as aggravation.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Number analyzed (Participants) | 129
participants
  Improvement | 122
  Aggravation | 7

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 30 days from the completion of assessments after the administration of the last study medication (follow-up) or the point of time of dropout
Description: Safety Population included all participants who took at least one dose of study drug.
Arm/Group | Osmotic Release Oral System (OROS) Methylphenidate HCL
Serious Adverse Events (participants affected / at risk) | 0/136
Other Adverse Events (participants affected / at risk) | 112/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osmotic Release Oral System (OROS) Methylphenidate HCL (N=136)
Insomnia (Psychiatric disorders) | 66
Anxiety (Psychiatric disorders) | 51
Decreased interest (Psychiatric disorders) | 41
Communication disorder (Psychiatric disorders) | 37
Onychophagia (Psychiatric disorders) | 37
Daydreaming (Psychiatric disorders) | 31
Nightmare (Psychiatric disorders) | 21
Depressed mood (Psychiatric disorders) | 18
Tic (Psychiatric disorders) | 11
Nervousness (Psychiatric disorders) | 9
Sleep disorder (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Hostility (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 2
Euphoric mood (Psychiatric disorders) | 2
Acute stress disorder (Psychiatric disorders) | 1
Logorrhoea (Psychiatric disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 82
Abdominal pain (Gastrointestinal disorders) | 43
Nausea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 41
Somnolence (Nervous system disorders) | 32
Dizziness (Nervous system disorders) | 19
Movement disorder (Nervous system disorders) | 3
Hypersomnia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Nasopharyngitis (Infections and infestations) | 11
Rhinitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Excessive eye blinking (Skin and subcutaneous tissue disorders) | 5
Eye pain (Skin and subcutaneous tissue disorders) | 1
Weight decreased (Investigations) | 4
Crying (General disorders) | 1
Inflammation (General disorders) | 1
Irritability (General disorders) | 1
Ear malformation (Congenital, familial and genetic disorders) | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1
Enuresis (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Depilation (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator cannot provide any trial related information to external parties' without mutual agreement with the sponsor. This is valid even after the contract is cancelled.